CLINICAL TRIAL: NCT02117999
Title: Randomized Clinical Trial Comparing Transepithelial Corneal Cross-linking Using Iontophoresis and Standard Corneal Cross-linking for the Treatment of Keratoconus
Brief Title: Transepithelial Corneal Cross-linking Using Iontophoresis
Acronym: T-iontoCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Collaborators: CNR Institute for chemical and physical processes (IPCF), Messina (Unknown)
Responsible Party: Principal Investigator, Marco Lombardo, Dr. Marco Lombardo, Fondazione G.B. Bietti, IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEA27; PON01_00110 (Other Grant/Funding Number: PON01_00110)
Record Dates: First submitted 2014-04-11; First posted 2014-04-21 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Progressive Keratoconus
Keywords: corneal cross-linking; transepithelial corneal cross-linking; iontophoresis; progressive keratoconus
MeSH Terms: interventions — Iontophoresis

STUDY DESIGN:
Intervention Model Description: Consecutive patients were randomized, using block randomization model, in one of the arm
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cross-linking with iontophoresis (Experimental): Transepithelial cross-linking by using iontophoresis to administer riboflavin into the corneal stroma
  Interventions: Device: Cross-linking with iontophoresis
- Standard corneal cross-linking (Active Comparator): Standard corneal cross-linking includes de-epithelialization and stromal soaking by applying drops of riboflavin
  Interventions: Device: Standard corneal cross-linking

INTERVENTIONS:
Device: Cross-linking with iontophoresis — The procedure involves a constant current source and two electrodes. The active electrode is a bath tube, which includes a stainless steel grid, placed into the cup at a minimal distance from the cornea. The reservoir is filled with dextran-free, hypotonic riboflavin-5-phosphate solution. The generator applies a constant current of 1mA for a preset period of 5 min. After the riboflavin administration by iontophoresis, the cornea is irradiated using a UVA lamp of 10mW/cm2 for 9 minutes.
  Other Names: Ricrolin+
  Arms: Cross-linking with iontophoresis
Device: Standard corneal cross-linking — In the standard CL, the epithelium is mechanically removed. Then, a solution of riboflavin is instilled each minute for 30 minutes. Corneas are irradiated using a UVA lamp of 3mW/cm2 for 30 minutes.
  Other Names: Ricrolin
  Arms: Standard corneal cross-linking

SUMMARY:
The purpose of the present Randomized Clinical Trial (RCT) is to compare the efficacy and safety of transepithelial corneal cross-linking using iontophoresis (T-ionto CL) to treat progressive keratoconus in comparison with standard cross-linking (standard CL).

DETAILED DESCRIPTION:
Keratoconus is a progressive corneal ectatic disease causing visual impairment by inducing irregular astigmatism and corneal opacity. This disorder typically begins during the second decade of life and, in severe forms, may need a corneal transplantation. Corneal cross-linking with riboflavin and UV-A is a procedure intended to halt keratoconus progression. It generates additional chemical bonds between stromal proteins in order to stiffen the corneal tissue. Standard CL includes epithelial removal and stroma soaking with dextran-enriched 0.1% riboflavin solution for 30 minutes before being exposed to ultraviolet-A radiation using a 3mW/cm2 lamp for 30 minutes.

Epithelial debridement exposes the cornea to a risk of side effects, such as pain for the first two post-operative days, temporary loss of visual acuity during the first three months, and serious complications, such as infection and stromal opacity due to corneal scarring.

Iontophoresis is a non invasive technique in which a weak electric current is used to enhance the penetration of hypotonic 0.1% riboflavin-5-phosphate solution into the corneal stroma through the intact epithelium. After iontophoresis, the corneal tissue is irradiated using a 10 mW/cm2 for 9 minutes (T-ionto CL). From previous experimental work (Lombardo M. et al. JCRS 2014 and JCRS 2015), the investigators provided evidence that T-ionto CL increases the stiffness of human corneas with results almost comparable with standard CL. The new procedure holds the promise to be as effective as the standard procedure while minimizing all the related risks. It is object of the present clinical trial to randomize patients with progressive keratoconus to T-ionto CL and standard CL and compare efficacy and safety of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive keratoconus

Exclusion Criteria:

* Anterior corneal curvature steeper than 61 D;
* central corneal thickness <400 um
* corneal scarring;
* descemetocele;
* history of herpetic keratitis;
* Concomitant eye diseases;
* Inflammatory eye diseases;
* Glaucoma;
* Cataract;
* Pregnancy

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Lombardo, MD, PhD, Principal Investigator — Fondazione G.B. Bietti, IRCCS
Locations (1):
- Fondazione G.B. Bietti, IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
still investigating this study population up to 3 years after treatment

REFERENCES:
- [Background] Spoerl E, Huhle M, Seiler T. Induction of cross-links in corneal tissue. Exp Eye Res. 1998 Jan;66(1):97-103. doi: 10.1006/exer.1997.0410. PMID 9533835
- [Background] Hao J, Li SK, Liu CY, Kao WW. Electrically assisted delivery of macromolecules into the corneal epithelium. Exp Eye Res. 2009 Dec;89(6):934-41. doi: 10.1016/j.exer.2009.08.001. Epub 2009 Aug 12. PMID 19682448
- [Background] Eljarrat-Binstock E, Domb AJ. Iontophoresis: a non-invasive ocular drug delivery. J Control Release. 2006 Feb 21;110(3):479-89. doi: 10.1016/j.jconrel.2005.09.049. Epub 2005 Dec 15. PMID 16343678
- [Background] Bikbova G, Bikbov M. Transepithelial corneal collagen cross-linking by iontophoresis of riboflavin. Acta Ophthalmol. 2014 Feb;92(1):e30-4. doi: 10.1111/aos.12235. Epub 2013 Jul 15. PMID 23848196
- [Background] Meek KM, Hayes S. Corneal cross-linking--a review. Ophthalmic Physiol Opt. 2013 Mar;33(2):78-93. doi: 10.1111/opo.12032. PMID 23406488
- [Derived] Lombardo M, Serrao S, Lombardo G, Schiano-Lomoriello D. Two-year outcomes of a randomized controlled trial of transepithelial corneal crosslinking with iontophoresis for keratoconus. J Cataract Refract Surg. 2019 Jul;45(7):992-1000. doi: 10.1016/j.jcrs.2019.01.026. Epub 2019 Apr 16. PMID 31003798
- [Derived] Lombardo M, Giannini D, Lombardo G, Serrao S. Randomized Controlled Trial Comparing Transepithelial Corneal Cross-linking Using Iontophoresis with the Dresden Protocol in Progressive Keratoconus. Ophthalmology. 2017 Jun;124(6):804-812. doi: 10.1016/j.ophtha.2017.01.040. Epub 2017 Mar 7. PMID 28283279
- See also: Inclusion and exclusion criteria to the present RCT are shown in the main website page — http://www.fondazionebietti.it

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were randomized after enrolment, with allocation ratio of 2:1, into either the study or control group
Pre-assignment Details: Block randomization strategy was used to randomize units with comparable baseline Kmax values in either group.
Units Other Than Participants: eyes
Groups:
- T-ionto CL: Eyes undergoing transepithelial corneal cross-linking with iontophoresis
- Standard CL: Eyes undergoing standard corneal cross-linking
Period: Overall Study
Arm/Group | T-ionto CL | Standard CL
Started | 20; 22 eyes | 10; 12 eyes
Mean Kmax Change in Corneal Topography | 20; 22 eyes | 10; 12 eyes
Completed | 20; 22 eyes | 10; 12 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Standard CL: Participants undergoing standard corneal cross-linking
- T-ionto CL: Participants undergoing transepithelial corneal cross-linking with iontophoresis
- Total: Total of all reporting groups
Arm/Group | Standard CL | T-ionto CL | Total
Number analyzed (Participants) | 10 | 20 | 30
Number analyzed (eyes) | 12 | 22 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.6) | 31 (6.6) | 30 (6)
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 4 | 3 | 7
  Male | 8 | 19 | 27
Ethnicity (NIH/OMB) [Count of Units; unit: eyes]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 22 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 22 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: eyes]
  Italy | 12 | 22 | 34
family history of keratoconus [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: K-max
Description: Measuring maximum keratometry (K-max), measured in diopters (D), derived from computerized videokeratography.
Time Frame: Changes from baseline in Kmax at 12 months
Population: Analysis of changes from baseline in each group was made using the paired Student t-test. Treatment effects were assessed using repeated measures ANOVA between groups and time (3 days, 7 days, 1-, 3-, 6- and 12-months). The outcome measures over time were corrected for baseline values.
Measure: Mean (Standard Deviation); unit: Diopters (D)
Groups:
- Transepithelial Corneal Cross-linking Using Iontophoresis: Transepithelial corneal cross-linking using iontophoresis
  Transepithelial corneal cross-linking using iontophoresis: The procedure involves a constant current source and two electrodes. The active electrode is a bath tube, which includes a stainless steel grid, placed into the cup at a minimal distance from the cornea. The reservoir is filled with dextran-free, hypotonic riboflavin-5-phosphate solution. The generator applies a constant current of 1mA for a preset period of 5 min. After the riboflavin administration by iontophoresis, the cornea is irradiated using a UVA lamp of 10mW/cm2 for 9 minutes.
- Standard Corneal Cross-linking: Standard corneal cross-linking
  Standard corneal cross-linking: In the standard CL, the epithelium is mechanically removed. Then, a solution of riboflavin is instilled each minute for 30 minutes. Corneas are irradiated using a UVA lamp of 3mW/cm2 for 30 minutes.
Arm/Group | Transepithelial Corneal Cross-linking Using Iontophoresis | Standard Corneal Cross-linking
Number analyzed (Participants) | 22 | 12
Diopters (D) | -0.52 (1.30) | -0.82 (1.20)
Statistical Analysis 1: Comparison: Transepithelial Corneal Cross-linking Using Iontophoresis vs Standard Corneal Cross-linking; Analysis of changes from baseline in each group was made using the paired Student t-test. Treatment effects were assessed using repeated measures ANOVA between groups and time (3 days, 7 days, 1-, 3-, 6- and 12-months). The outcome measures over time were corrected for baseline values. The relationship between the change in Kmax at 12 months and baseline parameters was assessed using Pearson's correlation analysis for either group; Test type: Non-Inferiority — Sample size calculation was performed to detect a difference of 0.95 D between the average Kmax changes for the T-ionto CL and standard CL groups at 12 months, at a significance level of 5% and a power of 81%, assuming a standard deviation of 1.20 D; p < 0.05, ANOVA

2. Primary Outcome: Corneal Endothelial Cell Density
Description: Endothelial cell density (ECD) will be evaluated using specular microscopy
Time Frame: Changes from baseline in ECD at 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | Transepithelial Corneal Cross-linking Using Iontophoresis | Standard Corneal Cross-linking
Number analyzed (Participants) | 22 | 12
cells/mm2 | 2675 (311) | 2658 (321)
Statistical Analysis 1: Comparison: Transepithelial Corneal Cross-linking Using Iontophoresis vs Standard Corneal Cross-linking; Analysis of changes from baseline in each group was made using the paired Student t-test. Treatment effects were assessed using repeated measures ANOVA between groups and time (3 days, 7 days, 1-, 3-, 6- and 12-months). The outcome measures over time were corrected for baseline values; Test type: Non-Inferiority — sample size calculation was performed to detect a difference of 0.95 D between the average Kmax changes for the T-ionto CL and standard CL groups at 12 months, at a significance level of 5% and a power of 81%, assuming a standard deviation of 1.20 D. The sample size of the study was 34 cases (allocation ratio of 2:1); p = 0.05, ANOVA; Mean Difference (Final Values) = 35

3. Secondary Outcome: Optical Aberrations
Description: Optical aberrations of the eye will be measured using dynamic skyascopy. Corneal wavefront aberration will be measured using Placido disk topographer and Scheimpflug tomographer.
Time Frame: Changes from baseline at 12 months.
Population: Corneal high-order aberrations
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | T-ionto CL | Standard CL
Number analyzed (Participants) | 20 | 10
micrometers | 2.19 (0.99) | 2.21 (0.86)

4. Secondary Outcome: Visual Acuity
Description: Visual acuity tested using ETDRS
Time Frame: Changes from baseline at 12 months.
Population: Corrected distance visual acuity
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | T-ionto CL | Standard CL
Number analyzed (Participants) | 20 | 10
LogMAR | 0.03 (0.10) | 0.01 (0.10)

5. Secondary Outcome: Contrast Sensitivity
Description: Contrast sensitivity tested using Pelli-Robson chart
Time Frame: Changes from baseline at 12 months.
Population: Contrast-sensitivity function assessed by Pelli-Robson charts
Measure: Mean (Standard Deviation); unit: log
Arm/Group | T-ionto CL | Standard CL
Number analyzed (Participants) | 20 | 10
log | 1.62 (0.08) | 1.63 (0.06)

6. Secondary Outcome: Central Retinal Thickness
Description: Central retinal thickness (1 mm ETDRS map) will be measured before and after CXL procedures
Time Frame: Changes from baseline at 12 months.
Population: 1 mm central retinal thickness assessed by SD-OCT
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | T-ionto CL | Standard CL
Number analyzed (Participants) | 20 | 10
micrometers | 275 (20) | 277 (38)

ADVERSE EVENTS:
Time Frame: 1 year
Description: no differences
Groups:
- Transepithelial Corneal Cross-linking Using Iontophoresis: Participants undergoing transepithelial corneal cross-linking using iontophoresis
- Standard Corneal Cross-linking: Participants undergoing standard corneal cross-linking
Arm/Group | Transepithelial Corneal Cross-linking Using Iontophoresis | Standard Corneal Cross-linking
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transepithelial Corneal Cross-linking Using Iontophoresis (N=20) | Standard Corneal Cross-linking (N=10)
Corneal sub-epithelial infiltrates (Eye disorders) | 0 (0) | 1 (1) — Corneal peripheral sub-epithelial infiltrates

LIMITATIONS AND CAVEATS:
Principal Investigator (PI) is NOT employed by the organization sponsoring the study. There is NOT an agreement between the PI and the Sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No